CLINICAL TRIAL: NCT05224518
Title: National Taiwan University Hospital Hsin-Chu Branch.
Brief Title: Exercise Intervention to Improve Quality of Life in Patients With Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 110-146-E
Record Dates: First submitted 2021-12-12; First posted 2022-02-04 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Fatigue; Quality of Life
Keywords: elastic band training; colorectal cancer; exercises
MeSH Terms: conditions — Colorectal Neoplasms; Fatigue; Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home-based elastic band training group (Experimental): The interventional group received 12 weeks of home-based elastic band training, three days a week, with progressive, medium-intensity exercise.
  Interventions: Behavioral: elastic band training
- stretching exercises group (Active Comparator): The control group received home stretching exercises three days a week for 12 weeks.
  Interventions: Behavioral: elastic band training

INTERVENTIONS:
Behavioral: elastic band training — elastic band training include stretching exercises
  Other Names: stretching exercises

SUMMARY:
The purpose of this study was to explore the 12-week effectiveness of home exercise intervention for colorectal cancer patients in improving fatigue, sleep, muscle endurance, and quality of life.

A. Explore the effect of "12-week home exercise intervention" in improving the fatigue of colorectal cancer patients.

B. Explore the effect of "12-week home exercise intervention" in improving the sleep quality of patients with colorectal cancer.

C. Explore the effect of "12-week home exercise intervention" in improving the muscle endurance of patients with colorectal cancer.

D. Explore the effect of "12-week home exercise intervention" in improving the quality of life of colorectal cancer patients.

DETAILED DESCRIPTION:
The study was conducted at the colon and rectal outpatient departments. A randomized controlled trial design was adopted. The participants were divided into an interventional group and a conventional therapy control group based on block randomization in a 1:1 ratio. Data were collected when patients returned to the clinic.

ELIGIBILITY:
A. Inclusion criteria

1. Above the age of 20, with colorectal cancer pathological stage in situ, I, II, and III.
2. Coherent, with no mental abnormalities.
3. Able to read Mandarin or communicate in Mandarin and Taiwanese to complete the questionnaire.
4. Provided informed consent.
5. No physical disabilities.

B. Exclusion criteria

1. Acute inflammation of the limbs and joints.
2. Previous abdominal surgery within 3 months.
3. Symptomatic cardiovascular events.
4. Long-term anti-depressant drug use.
5. Unilateral restrictions of the upper or lower limbs.
6. History of medium- or high-intensity exercise for more than half a year.
7. Having colostoma or ileostoma.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life of cancer patients(EORTC QLQ-C30) | baseline
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life of cancer patients(EORTC QLQ-C30) | 1rd month after recruited
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life of cancer patients(EORTC QLQ-C30) | 2rd month after recruited
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life of cancer patients(EORTC QLQ-C30) | 3rd month after recruited
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life of cancer patients(EORTC QLQ-C30) | 6rd month after recruited
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life of cancer patients(EORTC QLQ-C30) | 12rd month after recruited
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life of cancer patients(EORTC QLQ-C30) | 24rd month after recruited
  This questionnaire measures the general quality of life of cancer patients. There are 30 questions in total, including questions on physical functioning (5 questions), role function (2 questions), emotional functioning (4 questions),and cognitive functioning (2 questions), as well as, overall quality of life and health status (2 questions). And common symptoms such as fatigue (3 questions), pain (2 questions), nausea and vomiting (2 questions), dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial problems (one question each).
Quality of life of cancer patients(EORTC QLQ-CR29) | baseline
  The acceptance conditions of this study exclude cases of stomy; therefore, there is no score for stomy. Among these 21 questions, only body image, anxiety, weight, and sex are functional scales, and all the others are symptomatic. The higher the score, the more serious the symptom.
Quality of life of cancer patients(EORTC QLQ-CR29) | 1rd month after recruited
  The acceptance conditions of this study exclude cases of stomy; therefore, there is no score for stomy. Among these 21 questions, only body image, anxiety, weight, and sex are functional scales, and all the others are symptomatic. The higher the score, the more serious the symptom.
Quality of life of cancer patients(EORTC QLQ-CR29) | 2rd month after recruited
  The acceptance conditions of this study exclude cases of stomy; therefore, there is no score for stomy. Among these 21 questions, only body image, anxiety, weight, and sex are functional scales, and all the others are symptomatic. The higher the score, the more serious the symptom.
Quality of life of cancer patients(EORTC QLQ-CR29) | 3rd month after recruited
  The acceptance conditions of this study exclude cases of stomy; therefore, there is no score for stomy. Among these 21 questions, only body image, anxiety, weight, and sex are functional scales, and all the others are symptomatic. The higher the score, the more serious the symptom.
Quality of life of cancer patients(EORTC QLQ-CR29) | 6rd month after recruited
  The acceptance conditions of this study exclude cases of stomy; therefore, there is no score for stomy. Among these 21 questions, only body image, anxiety, weight, and sex are functional scales, and all the others are symptomatic. The higher the score, the more serious the symptom.
Quality of life of cancer patients(EORTC QLQ-CR29) | 12rd month after recruited
  The acceptance conditions of this study exclude cases of stomy; therefore, there is no score for stomy. Among these 21 questions, only body image, anxiety, weight, and sex are functional scales, and all the others are symptomatic. The higher the score, the more serious the symptom.
Quality of life of cancer patients(EORTC QLQ-CR29) | 24rd month after recruited
  The acceptance conditions of this study exclude cases of stomy; therefore, there is no score for stomy. Among these 21 questions, only body image, anxiety, weight, and sex are functional scales, and all the others are symptomatic. The higher the score, the more serious the symptom.

SECONDARY OUTCOMES:
Brief Fatigue Inventory-Taiwanese (BFI-T) | baseline
  The Taiwanese Behavior Inventory (BFI-T) has nine questions. The content is divided into two parts: the first part uses three questions to describe the current, average, and most serious degree of fatigue that the patient has experienced, and the second part uses six questions to describe the intensity of the disturbance to life, general activities, emotions, walking ability, and normal work.
  An 11-Point Likert scale from 0-10 is used to measure fatigue. Briefly, 0 means no feature; 10 means the most serious feature; 1-4 points to distinguish; 5-6 points mean moderate intensity; and 7-9 means severe intensity. In measuring interference with life: 0 means no interference; 10 means complete interference; 1-4 points mean life interference intensity is mild; 5-6 points mean life interference intensity is moderate; and 7-9 points mean life interference intensity is severe.
Brief Fatigue Inventory-Taiwanese (BFI-T) | 1rd month after recruited
  The Taiwanese Behavior Inventory (BFI-T) has nine questions. The content is divided into two parts: the first part uses three questions to describe the current, average, and most serious degree of fatigue that the patient has experienced, and the second part uses six questions to describe the intensity of the disturbance to life, general activities, emotions, walking ability, and normal work.
  An 11-Point Likert scale from 0-10 is used to measure fatigue. Briefly, 0 means no feature; 10 means the most serious feature; 1-4 points to distinguish; 5-6 points mean moderate intensity; and 7-9 means severe intensity. In measuring interference with life: 0 means no interference; 10 means complete interference; 1-4 points mean life interference intensity is mild; 5-6 points mean life interference intensity is moderate; and 7-9 points mean life interference intensity is severe.
Brief Fatigue Inventory-Taiwanese (BFI-T) | 2rd month after recruited
  The Taiwanese Behavior Inventory (BFI-T) has nine questions. The content is divided into two parts: the first part uses three questions to describe the current, average, and most serious degree of fatigue that the patient has experienced, and the second part uses six questions to describe the intensity of the disturbance to life, general activities, emotions, walking ability, and normal work.
  An 11-Point Likert scale from 0-10 is used to measure fatigue. Briefly, 0 means no feature; 10 means the most serious feature; 1-4 points to distinguish; 5-6 points mean moderate intensity; and 7-9 means severe intensity. In measuring interference with life: 0 means no interference; 10 means complete interference; 1-4 points mean life interference intensity is mild; 5-6 points mean life interference intensity is moderate; and 7-9 points mean life interference intensity is severe.
Brief Fatigue Inventory-Taiwanese (BFI-T) | 3rd month after recruited
  The Taiwanese Behavior Inventory (BFI-T) has nine questions. The content is divided into two parts: the first part uses three questions to describe the current, average, and most serious degree of fatigue that the patient has experienced, and the second part uses six questions to describe the intensity of the disturbance to life, general activities, emotions, walking ability, and normal work.
  An 11-Point Likert scale from 0-10 is used to measure fatigue. Briefly, 0 means no feature; 10 means the most serious feature; 1-4 points to distinguish; 5-6 points mean moderate intensity; and 7-9 means severe intensity. In measuring interference with life: 0 means no interference; 10 means complete interference; 1-4 points mean life interference intensity is mild; 5-6 points mean life interference intensity is moderate; and 7-9 points mean life interference intensity is severe.
Brief Fatigue Inventory-Taiwanese (BFI-T) | 6rd month after recruited
  The Taiwanese Behavior Inventory (BFI-T) has nine questions. The content is divided into two parts: the first part uses three questions to describe the current, average, and most serious degree of fatigue that the patient has experienced, and the second part uses six questions to describe the intensity of the disturbance to life, general activities, emotions, walking ability, and normal work.
  An 11-Point Likert scale from 0-10 is used to measure fatigue. Briefly, 0 means no feature; 10 means the most serious feature; 1-4 points to distinguish; 5-6 points mean moderate intensity; and 7-9 means severe intensity. In measuring interference with life: 0 means no interference; 10 means complete interference; 1-4 points mean life interference intensity is mild; 5-6 points mean life interference intensity is moderate; and 7-9 points mean life interference intensity is severe.
Brief Fatigue Inventory-Taiwanese (BFI-T) | 12rd month after recruited
  The Taiwanese Behavior Inventory (BFI-T) has nine questions. The content is divided into two parts: the first part uses three questions to describe the current, average, and most serious degree of fatigue that the patient has experienced, and the second part uses six questions to describe the intensity of the disturbance to life, general activities, emotions, walking ability, and normal work.
  An 11-Point Likert scale from 0-10 is used to measure fatigue. Briefly, 0 means no feature; 10 means the most serious feature; 1-4 points to distinguish; 5-6 points mean moderate intensity; and 7-9 means severe intensity. In measuring interference with life: 0 means no interference; 10 means complete interference; 1-4 points mean life interference intensity is mild; 5-6 points mean life interference intensity is moderate; and 7-9 points mean life interference intensity is severe.
Brief Fatigue Inventory-Taiwanese (BFI-T) | 24rd month after recruited
  The Taiwanese Behavior Inventory (BFI-T) has nine questions. The content is divided into two parts: the first part uses three questions to describe the current, average, and most serious degree of fatigue that the patient has experienced, and the second part uses six questions to describe the intensity of the disturbance to life, general activities, emotions, walking ability, and normal work.
  An 11-Point Likert scale from 0-10 is used to measure fatigue. Briefly, 0 means no feature; 10 means the most serious feature; 1-4 points to distinguish; 5-6 points mean moderate intensity; and 7-9 means severe intensity. In measuring interference with life: 0 means no interference; 10 means complete interference; 1-4 points mean life interference intensity is mild; 5-6 points mean life interference intensity is moderate; and 7-9 points mean life interference intensity is severe.
Pittsburgh Sleep Quality Index (PSQI) | baseline
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sexual sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Pittsburgh Sleep Quality Index (PSQI) | 1rd month after recruited
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sexual sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Pittsburgh Sleep Quality Index (PSQI) | 2rd month after recruited
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sexual sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Pittsburgh Sleep Quality Index (PSQI) | 3rd month after recruited
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sexual sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Pittsburgh Sleep Quality Index (PSQI) | 6rd month after recruited
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sexual sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Pittsburgh Sleep Quality Index (PSQI) | 12rd month after recruited
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sexual sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
Pittsburgh Sleep Quality Index (PSQI) | 24rd month after recruited
  The scale consists of 19 questions covering collective sleep quality, sleep latency, total sleep hours, sexual sleep habits, sleep disturbance, use of sleeping drugs, and daytime functioning.
  The PSQI score is calculated from the above seven facets. The score of each facet was 0-3 points, and the total score was 0-21 points. A score greater than 5 indicates that the total quality of sleep is poor.
3-d Physical Activity Record, 3-dPAR | baseline
  Developed in 1983, this evaluation divides the day from 7 am to midnight into 15 minutes, and divides common activities into the following categories: eating, working, transportation, sleeping, bathing, sports activities, etc., the intensity of which is categorized as very light, light, medium, and strong, and the activity type is coded as level 1-9: corresponding to 1.0-7.8 metabolic equivalent of task (MET) or higher, so as to record three-day physical activity and evaluate the energy consumed and time spent on different activities.
3-d Physical Activity Record, 3-dPAR | 3rd month after recruited
  Developed in 1983, this evaluation divides the day from 7 am to midnight into 15 minutes, and divides common activities into the following categories: eating, working, transportation, sleeping, bathing, sports activities, etc., the intensity of which is categorized as very light, light, medium, and strong, and the activity type is coded as level 1-9: corresponding to 1.0-7.8 metabolic equivalent of task (MET) or higher, so as to record three-day physical activity and evaluate the energy consumed and time spent on different activities.
30-second Chair sit-to-stand, 30-s STS | baseline
  Ability to test mobility and posture transposition. Using a chair without armrests, the number of times the participant could change from a sitting state (leaning back on the chair with both feet on the ground) to fully standing within 30 s was counted. Two tests were performed, with 1 min of rest in between, and the average value was rounded to the nearest value.
30-second Chair sit-to-stand, 30-s STS | 3rd month after recruited
  Ability to test mobility and posture transposition. Using a chair without armrests, the number of times the participant could change from a sitting state (leaning back on the chair with both feet on the ground) to fully standing within 30 s was counted. Two tests were performed, with 1 min of rest in between, and the average value was rounded to the nearest value.
Six-Minute Walk Test, 6MWT | baseline
  Functional quantitative indicators for measuring athletic ability and endurance.
  The participant is asked to walk on a 30-meter flat, straight walkway, marked with red tape every 3 m, and the distance traveled by the individual in six minutes is measured.
Six-Minute Walk Test, 6MWT | 3rd month after recruited
  Functional quantitative indicators for measuring athletic ability and endurance.
  The participant is asked to walk on a 30-meter flat, straight walkway, marked with red tape every 3 m, and the distance traveled by the individual in six minutes is measured.
Exercise Counseling and Programming Preferences | baseline
  Exercise preferences were assessed by questions related to exercise counseling and exercise programming.
Exercise Counseling and Programming Preferences | 3rd month after recruited
  Exercise preferences were assessed by questions related to exercise counseling and exercise programming.
Exercise Counseling and Programming Preferences | 6rd month after recruited
  Exercise preferences were assessed by questions related to exercise counseling and exercise programming.
Exercise Counseling and Programming Preferences | 12rd month after recruited
  Exercise preferences were assessed by questions related to exercise counseling and exercise programming.
Exercise Counseling and Programming Preferences | 24rd month after recruited
  Exercise preferences were assessed by questions related to exercise counseling and exercise programming.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, Study Chair — University of Nursing and Health Sciences, Taipei, Taiwan
Locations (1):
- NTU Hsin-Chu Hospital, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 24 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and receive the authors consent.

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Chen Y, Niu M, Zhang X, Qian H, Xie A, Wang X. Effects of home-based lower limb resistance training on muscle strength and functional status in stable Chronic obstructive pulmonary disease patients. J Clin Nurs. 2018 Mar;27(5-6):e1022-e1037. doi: 10.1111/jocn.14131. Epub 2018 Feb 6. PMID 29076609
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Result] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Result] Patel AV, Friedenreich CM, Moore SC, Hayes SC, Silver JK, Campbell KL, Winters-Stone K, Gerber LH, George SM, Fulton JE, Denlinger C, Morris GS, Hue T, Schmitz KH, Matthews CE. American College of Sports Medicine Roundtable Report on Physical Activity, Sedentary Behavior, and Cancer Prevention and Control. Med Sci Sports Exerc. 2019 Nov;51(11):2391-2402. doi: 10.1249/MSS.0000000000002117. PMID 31626056
- [Result] Uster A, Ruehlin M, Mey S, Gisi D, Knols R, Imoberdorf R, Pless M, Ballmer PE. Effects of nutrition and physical exercise intervention in palliative cancer patients: A randomized controlled trial. Clin Nutr. 2018 Aug;37(4):1202-1209. doi: 10.1016/j.clnu.2017.05.027. Epub 2017 Jun 8. PMID 28651827
- See also: National cancer institute. — https://www.cancer.gov/about-cancer/treatment/side-effects/fatigue/fatigue-hp-pdq